CLINICAL TRIAL: NCT06523127
Title: Withholding of Life-sustaining Treatment and Quality of Life After Severe Acute Brain Injury: Qualitative Analysis and Ethical Issues.
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN672024/CHUSTE
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Quality of Life; Brain Injuries; Post ICU
Keywords: Quality of life; Withholding of life-sustaining treatments; Withdrawal of life-sustaining treatment; Severe acute brain injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with severe acute brain injury and with withholding of life-sustaining treatment: Assessment of quality of life in patients with severe acute brain injury based on the audio recording during post-ICU follow-up.
  Interventions: Other: Recording data from the ICU stay and the post-ICU follow-up.
- Patients with severe acute brain injury and without withholding of life-sustaining treatment: Assessment of quality of life in patients with severe acute brain injury based on the audio recording during post-ICU follow-up.
  Interventions: Other: Recording data from the ICU stay and the post-ICU follow-up.

INTERVENTIONS:
Other: Recording data from the ICU stay and the post-ICU follow-up. — Record analysis of the post-ICU follow-up with the Interpretative Phenomenological Analysis

SUMMARY:
Withdrawal of life-sustaining treatment affects 10-15% of ICU patients, including those with severe acute brain injury, whose care appears futile in terms of prognosis based on clinical and paraclinical data, expected quality of life, patient preferences, age, or reduced quality of life.

There are few studies on withholding treatment compared with withdrawing treatment, and even fewer on survivors after a decision to withhold treatment.

Quality of life is defined by WHO as "an individual's perception of his or her position in life in the context of the culture and value systems in which he or she lives and in relation to his or her goals, expectations, standards and concerns". The relationship between quality of life and neurological outcome after severe acute brain injury is controversial and therefore difficult to predict.

That's why the investigators question the legitimacy of making decisions to withhold treatment from patients with severe acute brain injury based on their expected quality of life, when this prediction is uncertain.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* with severe acute brain injury (TBI, stroke, central nervous system infection).
* admitted in the neurocritical care unit in 2022.
* followed up 24 months after ICU between 15th April 2024 and 31st August 2024.

Exclusion Criteria:

Patients:

* death in 2024,
* refusal by patient or relative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute brain injury admitted to intensive care in 2022 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Interpretative Phenomenological Analysis | 24 months after ICU discharge
  Qualitative analysis of the quality of life in patients with severe acute brain injury and with withholding of life-sustaining treatment

SECONDARY OUTCOMES:
International survey among neurointensivists from ANARLF network - questionnaires | Month : 3
  Comparison of the number of decisions of withholding treatment in the clinical cases versus real life
International survey among neurointensivists from ANARLF network - follow-up | Month : 3
  Comparison of the predicted neurological outcome and quality of life by neurointensivists versus the real neurological outcome and quality of life assessed at the post-ICU follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Marie DAKENG, resident, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No